CLINICAL TRIAL: NCT00389805
Title: Phase I/II Study of Two Different Schedules of Bortezomib (VELCADE, PS-341) and Pemetrexed (ALIMTA) in Advanced Solid Tumors, With Emphasis on Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Bortezomib and Pemetrexed Disodium in Treating Patients With Advanced Non-Small Cell Lung Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#158; 200412739 (Other: UC Davis); H3E-US-X038 (Other: Eli Lilly)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; Pemetrexed; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: bortezomib
Drug: pemetrexed disodium
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: flow cytometry
Other: immunoenzyme technique
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Bortezomib and pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bortezomib together with pemetrexed disodium may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of two different schedules of bortezomib when given together with pemetrexed disodium and to see how well they work in treating patients with advanced non-small cell lung cancer or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety, including dose-limiting toxicities, and feasibility of combining bortezomib with pemetrexed disodium in patients with advanced non-small cell lung cancer (NSCLC) or other solid tumors. (Phase I)
* Determine the response rate in patients with advanced NSCLC treated with this regimen. (Phase II)

Secondary

* Compare the toxicity of 2 different schedules of bortezomib and pemetrexed disodium in patients with advanced solid tumors. (Phase I)
* Determine the maximum tolerated dose (MTD) of bortezomib when administered with pemetrexed disodium in 2 different treatment schedules in these patients. (Phase I)
* Determine, preliminarily, the efficacy of the combination of bortezomib and pemetrexed disodium in patients with advanced solid tumors. (Phase I)
* Assess the overall survival and progression-free survival of these patients. (Phase II)
* Evaluate the frequency and severity of toxicities associated with this regimen. (Phase II)

Tertiary

* Perform laboratory correlative studies on tumor tissue and blood samples to investigate potential predictors of response. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of bortezomib followed by a phase II, open-label study.

* Phase I: Patients will be accrued, in an alternating fashion, to 1 of 2 treatment groups.

  * Group I: Patients receive pemetrexed disodium IV on day 1 and bortezomib IV on days 1, 4, 8, and 11.
  * Group II: Patients receive pemetrexed disodium IV on day 1 and bortezomib IV on days 1 and 8.

In both groups, treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients per group receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive pemetrexed disodium bortezomib (at the MTD) as in either group I or group II of the phase I portion of the study. Selection of the treatment schedule is based upon observed toxicity, safety, tolerability, efficacy, and clinical practicality.

Blood is drawn at baseline and prior to courses 2 and 3 for correlative and molecular studies.

Tumor tissue and blood samples from patients enrolled in the phase II portion of the study are examined for various biological markers. Immunohistochemistry is used to measure BCL-2 gene, BCL-xL gene, BAX gene, and p27. Reverse transcriptase-polymerase chain reaction is used to assay the expression of thymidylate synthase, folsyl-polyglutamate synthase, and reduced folate carrier. Levels of plasminogen-activator inhibitor 1 gene, vascular endothelial growth factor, and osteopontin are measured by immunoenzyme techniques. The nuclear expression of NF-kB and p27 in blood is compared before and after study treatment by flow cytometry.

After completion of study treatment, patients in phase I are followed for 30 days and patients in phase II are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed diagnosis of 1 of the following:

  * Advanced solid tumor that progressed after standard therapy or for which no effective curative therapy exists (phase I)
  * Stage IIIB (pleural effusion) or IV non-small cell lung cancer (NSCLC) (phase II)

    * Disease must have progressed or recurred after 1 platinum-based therapy regimen
    * NSCLC that has progressed or recurred after first-line therapy for stage IIIA or IIIB disease allowed
* Measurable disease

  * Disease in previously irradiated sites is considered measurable if there is clear disease progression following radiotherapy
  * Evaluable disease (bone metastases, pleural fluid, ascites) allowed (phase I)
* No symptomatic brain metastasis or disease requiring steroids and anticonvulsants

  * Asymptomatic, previously treated (surgical resection or radiotherapy) brain metastases allowed provided patient is neurologically stable and has been off steroids and anticonvulsants for ≥ 4 weeks

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2 (phase I) or 0-1 (phase II)
* Life expectancy ≥ 3 months
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* AST ≤ 2.5 times upper limit of normal
* Granulocyte count ≥ 1,500/mm³
* Platelet count of ≥ 100,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No pre-existing neuropathy ≥ grade 2
* No other prior malignancy except for the following (phase II):

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer currently in complete remission
  * Any other cancer from which the patient has been disease free for > 5 years
* No hypersensitivity to bortezomib, boron, or mannitol
* No cardiovascular complications, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Electrocardiographic (ECG) evidence of acute ischemia or active conduction system abnormalities

    * Any ECG abnormality at screening must be documented as not medically relevant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bortezomib or pemetrexed disodium
* Any number of prior chemotherapy regimens allowed (phase I)
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C) and recovered
* More than 2 weeks since prior radiotherapy and recovered
* No nonsteroidal anti-inflammatory drugs (NSAIDs) or salicylates 2 days prior and 2 days after (5 days pre and post for long-acting NSAIDs) administration of pemetrexed disodium
* No concurrent anticonvulsants that are metabolized by the cytochrome P450 pathway

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Davies AM, Ho C, Metzger AS, Beckett LA, Christensen S, Tanaka M, Lara PN, Lau DH, Gandara DR. Phase I study of two different schedules of bortezomib and pemetrexed in advanced solid tumors with emphasis on non-small cell lung cancer. J Thorac Oncol. 2007 Dec;2(12):1112-6. doi: 10.1097/JTO.0b013e31815ba7d0. PMID 18090584

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Pemetrexed on day 1 (500 -600 mg/m2 IV) and bortezomib twice weekly (0.7-1.3mg/m3) on days 1, 4, 8, and 11 every 21 days
- Arm B: Pemetrexed on day 1 (500 -600 mg/m2 IV) and bortezomib twice weekly (0.7-1.3mg/m2) on days 1 and 8 every 21 days
Period: Phase I
Arm/Group | Arm A | Arm B
Started | 15 | 12
Completed | 15 | 12
Not Completed | 0 | 0
Period: Phase II
Arm/Group | Arm A | Arm B
Started | 0 (The Phase II study was not conducted.) | 0 (The Phase II study was not conducted.)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Pemetrexed on day 1 and bortezomib days 1, 4, 8, and 11 every 21 days
- Arm B: Pemetrexed on day 1 and bortezomib days 1 and 8 every 21 days
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 79] | 59 [45 to 80] | 60 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a Dose-limiting Toxicity (Phase I)
Description: Grade 4 thrombocytopenia or grade 3 thrombocytopenia associated with bleeding, requirement for transfusion or lasting >7 days; febrile neutropenia; grade 3 neutropenia associated with infection; any other grade >/=3 non-hematologic toxicity considered by the investigator to be related to study drug.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
Participants | 3 | 0

2. Primary Outcome: Number of Participants Who Experience Adverse Events (Phase I)
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 (Phase I).
Time Frame: Throughout the entire study (up to 36 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
Participants | 15 | 12

3. Primary Outcome: Number of Patients With Grade ≥ 3 Toxicity (Phase I)
Description: Grade 3/4 toxicity occurring in a patient within 1 cycle.
Time Frame: First cycle of treatment (3 weeks)
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
participants
  Neutropenia | 12 | 1
  Anemia | 1 | 0
  Thrombocytopenia | 0 | 1
  Increased transaminases | 1 | 0
  Fatigue | 2 | 0

4. Primary Outcome: Number of Patients Who Responded to Study Treatment (Phase II)
Description: To determine the response rate of bortezomib in combination with pemetrexed in patients with advanced NSCLC. Response rate was assessed by CT scan. CT scans was performed at baseline and every two cycles (prior to 3rd and 5th cycle). The evaluation of response was based on standard RECIST criteria.
Time Frame: From start of treatment until disease progression/recurrence.
Population: The Phase II study was not conducted.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients With Toxicity by NCI CTC v3.0 (Phase I)
Description: Adverse events possibly related to treatment, graded according to the NCI CTCAE v3.0.
Time Frame: Up to 36 months
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
participants
  Neutropenia | 12 | 1
  Anemia | 1 | 0
  Thrombocytopenia | 0 | 1
  Increased transaminases | 12 | 5
  Anorexia | 4 | 6
  Constipation | 5 | 3
  Cough | 5 | 4
  Dehydration | 4 | 1
  Diarrhea | 2 | 3
  Dizziness | 5 | 4
  Edema | 4 | 4
  Fatigue | 15 | 11
  Fever | 3 | 3
  Infection | 6 | 4
  Nausea +/- vomiting | 10 | 6
  Neuropathy | 4 | 6
  Rash | 6 | 5
  Renal impairment | 5 | 1
  Weakness | 0 | 2

6. Secondary Outcome: Maximum Tolerated Dose of Bortezomib in Combination With Pemetrexel (Phase I)
Time Frame: Up to 36 months
Measure: Number; unit: Mg/m^2
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
Mg/m^2 | 1.3 | 1.6

7. Secondary Outcome: Number of Participants With Response to Therapy as Measured by RECIST (Phase I)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Best overall response is the best response recorded from the start of the treatment until disease progression/recurrence.
Time Frame: Up to 36 months
Population: All patients for whom response evaluation measurements were recorded at baseline and after 2 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 12
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1 | 1
  Stable Disease (SD) | 7 | 6
  Progressive Disease (PD) | 7 | 5

8. Secondary Outcome: Number of Participants With Toxicities (Phase II)
Description: Each adverse event will be determined by using the NCI CTCAE, Version 3.0.
Time Frame: Up to 36 months
Population: The Phase II study was not conducted.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Analysis of Molecular Determinants in Tumor Samples (Phase II)
Description: Expression of relevant molecular targets of the proteasome, which is inhibited by bortezomib.
Time Frame: Up to 36 months
Population: The Phase II study was not conducted.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Importance of Folate-associated Gene Expression and Response or Outcome (Phase II)
Description: Overexpression of reduced folate carrier (RFC) protein is thought to contribute to decreased resistance to pemetrexed. Levels of expression will be studied by measuring mRNA transcripts using quantitative Reverse Transcriptase-Polymerase Chain Reaction in archival patient tumor specimens.
Time Frame: Up to 36 months
Population: The Phase II study was not conducted.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Effect of Bortezomib on Over Expression of NF-kB, BCL-2, and BCL-xL (Phase II)
Description: Tumor levels of BCL-2, BCL-xL and BAX will be assessed by immunohistochemistry (IHC).
Time Frame: Up to 36 months
Population: The Phase II study was not conducted.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 15/15 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=15) | Arm B (N=12)
Increased transaminases (Hepatobiliary disorders) | 12 | 5
Anorexia (Metabolism and nutrition disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dizziness (Nervous system disorders) | 5 | 4
Edema (General disorders) | 4 | 4
Fatigue (General disorders) | 15 | 11
Fever (General disorders) | 3 | 3
Infection (Infections and infestations) | 6 | 4
Nausea +/- vomiting (Gastrointestinal disorders) | 10 | 6
Neuropathy (Nervous system disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Renal impairment (Renal and urinary disorders) | 5 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 12 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes